CLINICAL TRIAL: NCT03477435
Title: Comparing an Opt-out to an opt-in Approach for Smoking Cessation in VA Primary Care Clinics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 17-056
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Use
Keywords: smoking; tobacco dependence; quitline; smoking cessation
MeSH Terms: conditions — Tobacco Use; Smoking; Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Type 1 hybrid effectiveness/implementation study to evaluate two population-based approaches
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opt-in clinical reminder (Experimental): As the investigators have done previously, the reminder will be self-explanatory, and will walk staff through each step of referral. The reminder will include the following domains: normative advice, referral to treatment, handout
  Interventions: Behavioral: Staff training and academic detailing
- Opt-out tobacco treatment (Experimental): The investigators will directly change the treatment status quo by implementing a clinical reminder that automatically initiates tobacco treatment referral at the time the reminder is activated.
  Interventions: Behavioral: Staff training and academic detailing

INTERVENTIONS:
Behavioral: Staff training and academic detailing — Both arms will receive training at baseline to help their patients quit smoking. The training will be a mix of content and process education. We will provide brief updates to staff every 6 months throughout the intervention period, which will focus primarily on process education. We will monitor which staff attend and reach out separately to staff who did not. During the month after implementation of the clinical reminders, two study investigators will make a brief outreach visit to each staff member. We will follow a script, using the seven steps recommended by the National Resource Center for Academic Detailing: 1) Introduction; 2) Needs Assessment; 3) Key Messages/Features/Benefits; 4) Understanding Barriers and Enablers; 5) Identifying and Handling Objections; 6) Summary; and 7) Close. The key message (Step 3) will include demonstration of the clinical reminder, review of the evidence for telephone counseling and text messaging and how to refer patients.

SUMMARY:
The investigators propose a Type I hybrid effectiveness/implementation study to evaluate two population-based approaches for increasing use of Quitlines and text messaging at two VA sites. Specifically, the investigators will test the default bias, examining whether an opt-out approach to referral is more effective than an opt-in approach. The investigators will randomly assign teams to either an opt-out or opt-in approach to referring smokers to treatment. In the opt-out approach, the default is that everyone is referred to treatment unless they actively choose not to be. In the opt-in approach, people are offered treatment but must actively choose to enroll in it.

DETAILED DESCRIPTION:
This project is a Type 1 hybrid effectiveness/implementation study to evaluate two population-based approaches for increasing use of specific evidence-based approaches for behavioral tobacco dependence treatment, Quitlines and text messaging, at the Manhattan and Brooklyn campuses of the VA New York Harbor Healthcare System (NYHHS). The project will test the default bias, examining whether an opt-out approach to referral is more effective than an opt-in approach. Researchers will randomly assign clinical care teams at each VA campus to either an opt-out or an opt-in approach to referring smokers to treatment. In the opt-out approach, the default is that everyone is referred to treatment unless they actively choose not to be. In the opt-in approach, people are offered treatment but must actively choose to enroll in it.

ELIGIBILITY:
Inclusion Criteria:

* Survey Cohort -- Have been seen by an NA on the PACT team in the past 12 months at the Manhattan or Brooklyn VA campus AND Current smoker
* Nursing Assistants/Registered Nurses -- Work on a PACT at the Manhattan or Brooklyn VA campus
* Administrative Cohort -- Have been seen by a PACT team at the Manhattan or Brooklyn VA campus AND Current smoker
* Patient Post-Visit Survey Population -- Had a visit with an NA/RN included in the study AND Current smoker

Exclusion Criteria:

* Survey Cohort -- Non-English speaking
* Nursing Assistants/Registered Nurses -- None
* Administrative Cohort -- None
* Patient Post-Visit Survey Population -- Non-English speaking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1365 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of smokers who accept referral to treatment (Quitline or text messaging) | 2-year intervention period
  This outcome will be based on intervention process data. Note that we will measure both offering and accepting referral, but our outcome will be accepting referral.
Proportion of smokers who engage in treatment with the Quitline or text messaging service | 2-year intervention period
  This outcome will be based on data from the Quitline and SmokefreeTXT.
Abstinence at the end of the 2-year intervention period | 7-day abstinence
  Abstinence will be based on self-report, as is recommended for population-level studies

SECONDARY OUTCOMES:
Cost-effectiveness of the two approaches (opt-out vs opt-in) | 2-year intervention period
  This outcome will be based on cost data at the end of the intervention
Use of smoking cessation medications | 2-year intervention period
  This outcome will be based on VA administrative data

CONTACTS AND LOCATIONS:
Overall Officials: Scott E. Sherman, MD MPH, Principal Investigator — VA NY Harbor Healthcare System, New York, NY; Steven S. Fu, MD MSCE, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haber Y, Fu SS, Rogers E, Richter K, Tenner C, Dognin J, Goldfeld K, Gold HT, Sherman SE. A novel opt-in vs opt-out approach to referral-based treatment of tobacco use in Veterans Affairs (VA) primary care clinics: A provider-level randomized controlled trial protocol. Contemp Clin Trials. 2022 May;116:106716. doi: 10.1016/j.cct.2022.106716. Epub 2022 Mar 8. PMID 35276337